CLINICAL TRIAL: NCT03177577
Title: Strengthening of the First Dorsal Interosseous for Thumb Carpometacarpal Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P002710
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Thumb Osteoarthritis; First Dorsal Interosseous Strengthening
MeSH Terms: interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Splint Only (Placebo Comparator): Subjects with carpometacarpal (CMC) osteoarthritis treated by splinting of their thumb.
  Interventions: Device: Splint
- Splint with first dorsal interosseous (FDI) strengthening (Active Comparator): Subjects with carpometacarpal (CMC) osteoarthritis treated by splinting of their thumb combined with first dorsal interosseous (FDI) strengthening stabilization exercises.
  Interventions: Device: Splint with strengthening exercises

INTERVENTIONS:
Device: Splint — Subjects will use a splint custom-made by Massachusetts General Hospital Occupational Therapists as part of standard care for treatment of carpometacarpal (CMC) osteoarthritis.
  Arms: Splint Only
Device: Splint with strengthening exercises — Subjects will use a splint custom-made by Massachusetts General Hospital Occupational Therapists as part of standard care for treatment of carpometacarpal (CMC) osteoarthritis and will also be taught two first dorsal interosseous (FDI) strengthening exercises.
  Arms: Splint with first dorsal interosseous (FDI) strengthening

SUMMARY:
To determine the effect of first dorsal interosseus (FDI) strengthening in patients with thumb carpometacarpal (CMC) osteoarthritis.

DETAILED DESCRIPTION:
Thumb CMC osteoarthritis is a normal part of aging. Most patients are able to adapt to symptoms of pain and disability, other patients might benefit from non-operative interventions; e.g. splinting, corticosteroid injections, pain medication, and multiple hand exercises.

The dorsal ligament complex is one of the components for stability of the thumb CMC joint. These ligaments specifically create stability for pinch and grip during the final phase of opposition. Both, the opponens pollicis (OP) and the first dorsal interosseous (FDI) play a key role in centralizing the metacarpal on the trapezium. A retrospective study showed that a dynamic stability modeled approach, including targeting the FDI, reduced pain and improved function in patients with thumb CMC osteoarthritis. Recently, another study demonstrated that reduction of radial subluxation - the thumb metacarpal versus the trapezium CMC joint - was achieved by contraction of the dynamic stabilizers of the healthy hand, specifically with the focus on the FDI.

More clinical research is needed to determine if there are efficacious (effective and low-cost) evidence-based exercise programs for pain reduction and functional improvement in patients with thumb CMC osteoarthritis. The investigators are interested in the effect of FDI strengthening in patients with thumb CMC osteoarthritis. Therefore, the investigators hypothesized that there is no difference in the change of lateral pinch strength at 12 weeks between patients treated with a splint versus patients treated with a splint and FDI strengthening for thumb CMC osteoarthritis. We also tested the same hypothesis for 3-point chuck strength, VAS for pain, and PROMIS Upper Extremity CAT.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* English-speaking
* Splint treatment for thumb carpometacarpal (CMC) osteoarthritis

Exclusion Criteria:

* Less than 18 years old
* Rheumatoid Arthritis or post-traumatic carpometacarpal (CMC) osteoarthritis
* Patients that received a corticosteroid injection during the appointment for treatment of thumb carpometacarpal (CMC) osteoarthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2025-06 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Difference in 3-point chuck strength at 12 weeks | At enrollment and 12 week follow up
  Investigators will measure the pinch strength by placing a pinch meter between the pad of the thumb and pad of the index and middle finger. The investigators will compare the change in 3 point chuck strength between the two cohorts after 12 weeks of treatment.
Difference in Lateral pinch strength at 12 weeks | At enrollment and 12 week follow up
  The investigators will measure lateral pinch strength by placing a pinch meter between the pad of the thumb and lateral surface of the index finger. The investigators will compare the change in lateral pinch strength between the two cohorts after 12 weeks of treatment.
Visual Analog Scale (VAS) for Pain | At enrollment and 12 week follow up
  The Visual Analog Scale for Pain measures the amount of pain on a scale from 0, no pain, to 10, worst possible pain. The investigators will compare the change in pain between the two cohorts after 12 weeks of treatment.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Upper Extremity Computer Adaptive Test (CAT) at 12 weeks | At Enrollment and 12 week follow up
  A computerized assessment of depression measured at enrollment. The average T score of the U.S. population is 50, so the T score reported compares the study population to the U.S. population, where a T score greater than 50 is worse than the average and a T score less than 50 is better than the average. The investigators will compare the change in PROMIS Upper Extremity between the two cohorts after 12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sodha S, Ring D, Zurakowski D, Jupiter JB. Prevalence of osteoarthrosis of the trapeziometacarpal joint. J Bone Joint Surg Am. 2005 Dec;87(12):2614-2618. doi: 10.2106/JBJS.E.00104. PMID 16322609
- [Background] Edmunds JO. Traumatic dislocations and instability of the trapeziometacarpal joint of the thumb. Hand Clin. 2006 Aug;22(3):365-92. doi: 10.1016/j.hcl.2006.05.001. PMID 16843802
- [Background] O'Brien VH, Giveans MR. Effects of a dynamic stability approach in conservative intervention of the carpometacarpal joint of the thumb: a retrospective study. J Hand Ther. 2013 Jan-Mar;26(1):44-51; quiz 52. doi: 10.1016/j.jht.2012.10.005. Epub 2012 Nov 21. PMID 23177671
- [Background] McGee C, O'Brien V, Van Nortwick S, Adams J, Van Heest A. First dorsal interosseous muscle contraction results in radiographic reduction of healthy thumb carpometacarpal joint. J Hand Ther. 2015 Oct-Dec;28(4):375-80; quiz 381. doi: 10.1016/j.jht.2015.06.002. Epub 2015 Jun 27. PMID 26209165